CLINICAL TRIAL: NCT05565950
Title: A Phase 1/2 Study to Establish An Initial Therapeutic Range and Safety Data for AI-09 in the Treatment of Glabellar Lines
Brief Title: AI-09 In Subjects With Glabellar Lines, GL-101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eirion Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: AI-09-GL-101
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Glabellar Frown Lines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (14):
- AI-09 Dose 1 (Experimental): Dose 1 of botulinum toxin, Type A, intramuscular injection, administered once at baseline
  Interventions: Biological: AI-09
- Vehicle Dose 1 (Placebo Comparator): Vehicle, intramuscular injection, administered once at baseline
  Interventions: Biological: Vehicle
- AI-09 Dose 2 (Experimental): Dose 2 of botulinum toxin, Type A, intra-muscular injection, administered once at baseline
  Interventions: Biological: AI-09
- Vehicle Dose 2 (Placebo Comparator): Vehicle, intramuscular injection, administered once at baseline
  Interventions: Biological: Vehicle
- AI-09 Dose 3 (Experimental): Dose 3 of botulinum toxin, Type A, intra-muscular injection, administered once at baseline
  Interventions: Biological: AI-09
- Vehicle Dose 3 (Placebo Comparator): Vehicle, intramuscular injection, administered once at baseline
  Interventions: Biological: Vehicle
- AI-09 Dose 4 (Experimental): Dose 4 of botulinum toxin, Type A, intra-muscular injection, administered once at baseline
  Interventions: Biological: AI-09
- Vehicle Dose 4 (Placebo Comparator): Vehicle, intramuscular injection, administered once at baseline
  Interventions: Biological: Vehicle
- AI-09 Dose 5 (Experimental): Dose 5 of botulinum toxin, Type A, intra-muscular injection, administered once at baseline
  Interventions: Biological: AI-09
- Vehicle Dose 5 (Placebo Comparator): Vehicle, intramuscular injection, administered once at baseline
  Interventions: Biological: Vehicle
- AI-09 Dose 6 (Experimental): Dose 6 of botulinum toxin, Type A, intra-muscular injection, administered once at baseline
  Interventions: Biological: AI-09
- Vehicle Dose 6 (Placebo Comparator): Vehicle, intramuscular injection, administered once at baseline
  Interventions: Biological: Vehicle
- AI-09 Dose 7 (Experimental): Dose 7 of botulinum toxin, Type A, intra-muscular injection, administered once at baseline
  Interventions: Biological: AI-09
- Vehicle Dose 7 (Placebo Comparator): Vehicle, intramuscular injection, administered once at baseline
  Interventions: Biological: Vehicle

INTERVENTIONS:
Biological: AI-09 — Botulinum toxin, Type A, intramuscular injection, administered once at baseline
  Arms: AI-09 Dose 1; AI-09 Dose 2; AI-09 Dose 3; AI-09 Dose 4; AI-09 Dose 5; AI-09 Dose 6; AI-09 Dose 7
Biological: Vehicle — Vehicle Formulation
  Arms: Vehicle Dose 1; Vehicle Dose 2; Vehicle Dose 3; Vehicle Dose 4; Vehicle Dose 5; Vehicle Dose 6; Vehicle Dose 7

SUMMARY:
AI-09 In Subjects with Glabellar Lines

DETAILED DESCRIPTION:
A Phase 1/2, multicenter, out-patient, prospectively randomized, double-blind, vehicle-controlled study to establish an initial therapeutic range for AI-09 in the treatment of glabellar lines and provide initial data regarding its potential safety.

ELIGIBILITY:
Inclusion Criteria:

* able to understand and give written informed consent
* willingness to have their pictures taken
* 20 - 70 years of age
* moderate to severe glabellar lines (IGA 2-3) on contraction
* moderate to severe glabellar lines (SSA 2-3) on contraction
* none to mild glabellar lines wrinkles (IGA 0-1) at rest
* willingness to refrain from the use of facial fillers, retinoids, Botox, laser treatments, or any product affecting skin remodeling or that might cause an active dermal response during the course of the study
* female subjects of child-bearing potential must have a negative urine pregnancy test and be non-lactating at the Baseline visit
* female subjects of child-bearing potential must utilize one of the following methods of birth control throughout the study: IUD, diaphragm, a condom, a spermicidal gel or foam, oral contraceptives (provided subject has been utilizing this method for at least 4 months prior to Baseline and has not changed the brand within this period), or patch, injectable, implantable, or vaginal ring contraceptives. Subjects may also participate if they are surgically sterilized (tubal sterilization or hysterectomy)
* subjects should be in good general health as determined by the investigator and free of any disease that may interfere with study evaluations or the Investigational Product

Exclusion Criteria:

* the inability to substantially lessen glabellar lines by physically spreading them apart
* excessive weakness or atrophy in the target muscle(s)
* eyelid ptosis
* presence or history of "dry eye"
* history of periocular surgery, brow lift or related procedures, or deep dermal scarring
* concurrent or recent (within the last 6 months) use of any other botulinum toxin drug product anywhere in the body
* history of immunization or hypersensitivity to any botulinum toxin serotype
* history of non-response to any prior botulinum toxin treatments
* anticipated need for treatment with botulinum toxin of any serotype for a reason during the trial (other than the investigational treatment)
* any medical condition that may put the subject at increased risk with exposure to botulinum toxin including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function
* pregnancy or lactation
* application of any topical prescription medication to the treatment area within 14 days prior to treatment
* subjects on clinically significant, concomitant drug therapy
* participation in another investigational drug trial or receiving any investigational treatment(s) within 30 days of Baseline
* alcohol or drug abuse within the past 3 years
* psychiatric disease interfering with the subject's ability to give informed consent
* refusal or inability to comply with the requirements of the protocol for any reason

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Investigators Global Assessment (IGA) | 18 Weeks (26 Weeks for Cohorts 4, 5 & 6)
  Investigators Global Assessment. Glabellar Line Severity scale where severity is scored between 0-4 (0=absent; 4=severe).

SECONDARY OUTCOMES:
Total Number of Observations With a Response Defined as Change ≥2 in IGA-C and SSA-C Score | Week 1, 2, 4, 8, 12, 18 (Week 26 assessments for Cohorts 4, 5 & 6)
  Total number of observations with a change in the Investigators Global Assessment on Contraction, IGA-C, and the Subject Self-Assessment on Contraction, SSA-C, using the Glabellar Line Severity scale (GLS), where severity is scored between 0-4 (0=absent; 4=severe). To count, a "responder" is defined as a change by at least two ordinals in both assessments.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Eirion Research Site, Boca Raton, Florida
  - Eirion Research Site, Miami, Florida

IPD SHARING:
Plan to Share IPD: No